CLINICAL TRIAL: NCT04602377
Title: Multicentric Non-randomized Phase II of Pembrolizumab in Combination With Etoposide-cisplatin-based Chemotherapy in First-line Small Cell Ovarian Carcinoma of Hypercalcemic Type
Brief Title: Addition of Pembrolizumab to the Standard of Care Chemotherapy in Patient With SCCOHT
Acronym: PembroSCCOHT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GINECO-OV243b
Record Dates: First submitted 2020-10-06; First posted 2020-10-26 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Small Cell Ovarian Carcinoma
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Single arm study
  Interventions: Drug: Pembrolizumab 25 MG/ML [Keytruda]

INTERVENTIONS:
Drug: Pembrolizumab 25 MG/ML [Keytruda] — Pembrolizumab (200mg flat dose) will be administred in combinaison with PAVEP chemotherapy for the first 6 cycles (21-day cycle)
  Then, Pembrolizumab (200mg flat dose) will be administred in monotherapy until one year for patients with complete response and up to two years for patients with Stable disease or Progression response after the end of first-sequence therapy (PAVEP chemotherapy +/- High dose chemotherapy) or until disease progression.
  Other Names: MK-3475

SUMMARY:
Small cell ovarian carcinomas are rare and have a very poor prognosis affecting a young population. The objective of this study is to increase the efficacy of the initial chemotherapy by providing immunotherapy and to be able to offer to more patients the possibility of benefiting from an intensification of chemotherapy, which is a major prognostic factor in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who are at least 12 years of age on the day of signing informed consent with previously untreated, pathologically confirmed Small cell carcinoma of the ovary.Patients could be included after one cycle of chemotherapy but have to start treatment within 4 weeks after the first cycle of chemotherapy. They will start the scheme at cycle 2.
2. Stage FIGO I to IV classification
3. Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
4. Have adequate organ function:

   * Adequate marrow function

     * White blood cell (WBC) >2000/mm3 (stable off any growth factor within 4 weeks of first study drug administration)
     * Neutrophils >1500/ mm3 (stable off any growth factor within 4 weeks of first study drug administration)
     * Platelets > 100 × 103/mm3 (transfusion to achieve this level is not permitted within 2 weeks of first study drug administration)
     * Haemoglobin > 9 g/dL (transfusion to achieve this level is not permitted within 2 weeks of first study drug administration)
   * Adequate other organ functions

     * ALT and AST < 3× institutional ULN
     * Total bilirubin < 1.5× institutional ULN (except Gilbert Syndrome: < 3.0 mg/dL)
     * Normal thyroid function, subclinical hypothyroidism (thyroid-stimulating hormone [TSH] < 10 mIU/mL) or have controlled hypothyroidism on appropriate thyroid supplementation
     * Left ventricular ejection fraction (LVEF) > 55 % measured by ECHO (preferred) or MUGA scans
     * Serum creatinine < 2× ULN or creatinine clearance (CrCl) > 60 mL/min (measured using the Cockcroft-Gault formula below):
5. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial, prior to any study-specific procedure. The participant may also provide consent for (140 - age in years) × weight in kg × 0.85 Female CrCl = 72 × serum creatinine in mg/dL GINECO-OV243b - PembroSCCOHT - Protocol - Version 1.2 - 10/09/2020 Page 7 sur 83 Future Biomedical Research. However, participant may participate in the main trial without participating in Future Biomedical Research.
6. Covered by a medical insurance
7. Stated willingness to comply with all study procedures and availability for the duration of the study
8. Women of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to treatment allocation
9. For females of reproductive potential: use of highly effective contraception throughout the study period up to 120 days after the last dose of pembrolizumab and 180 days following the end of chemoradiotherapy (if applicable).

Exclusion Criteria:

1. Prior therapy for the disease with chemotherapy and/or an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
2. Patients who have received a live vaccine within 30 days prior to the first dose of study drug.

   Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed. Inactivated rabies vaccines are allowed.
3. Patients who have had an allogenic tissue/solid organ transplant.
4. Patient who has received more than one cycle of platinum-based chemotherapy, or any prior systemic anti-cancer therapy including investigational agents for the SCCOHT. (Patients could be included after one cycle of platinum-based therapy).
5. Patients who have a known diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg prednisone daily or equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug.
6. Patients who have a known additional malignancy that is progressing or has required active treatment within the past 5 years.

   Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
7. Patients who have a contraindication to any component of cisplatin, adriamycine, vepeside and cyclophosphamide.

   Note: Investigators must use the local label for contraindications, prohibited medications, and precautions for use.
8. Patients who have severe hypersensitivity (Grade 3 or higher) to pembrolizumab and/or any of its excipients (refer to the IB for a list of excipients).
9. Patients who have a known severe hypersensitivity (Grade 3 or higher) to any of the study chemotherapy agents and/or to any of their excipients (refer to the approved product label(s) for a list of excipients).
10. Patients who have an active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
11. Patients who have a history of (non-infectious) pneumonitis/ interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease that requires steroids.
12. Has an active infection requiring systemic therapy.
13. Has a known history of human immunodeficiency virus (HIV) infection. HIV testing is not required unless mandated by local health authority.
14. Has a history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or active hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
15. Has a known history of active tuberculosis (TB; Bacillus tuberculosis)
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
17. Has a known psychiatric or substance abuse disorder that would interfere with cooperating with the requirements of the study.
18. Breastfeeding women
19. Participation in another clinical study with an investigational product 30 days prior and during the treatment course, and 30 days after end of treatment.

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-08-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | Around 4 to 6 months of the last patient included
  CRR is defined as the proportion of patients who reached complete response (CR), according to RECIST v1.1 after the first sequence therapy including chemotherapy associated with immunotherapy and surgery.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability of pembrolizumab in combinaison with chemotherapy] | 30 days after the end of Cycle 6 (each cycle is 21 days)
  Adverse Events will be described in terms of frequency according to CTCAE v5 grade
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability of pembrolizumab in monotherapy] | 30 days after last treatment intake
  Adverse Events will be described in terms of frequency according to CTCAE v5 grade
Progression Free Survival (PFS) | from date of inclusion to date of event, assessed up to 5 years
  PFS is defined as the time from inclusion until the date of event defined as the first objective documented progression, according to investigator assessment of RECIST v1.1 or death (by any cause in the absence of progression).
Overall Survival (OS) | from date of inclusion to death, assessed up to 5 years
  OS is defined as the time from the date of inclusion until death due to any cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.
Partial Response Rate (PRR) | Around 4 to 6 months of the last patient included
  PRR is defined as the proportion of patients who reached partial response (PR), at the end of first-sequence therapy, according to RECIST v1.1.
Duration of Response (DoR) | assessed up to 42 months
  DOR is defined as the duration from complete response is first met until the first objective documented progression, according to RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia PAUTIER, MD, PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (13):
- France (13):
  - ICO - Paul Papin, Angers
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Centre Hospitalier Régional Universitaire de Besançon, Besançon
  - Institut Bergonié, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - ICM Val d'Aurelle, Montpellier
  - ICANS - Institut de cancérologie Strasbourg Europe, Strasbourg
  - Hôpital de Hautepierre, Strasbourg
  - Oncopole Claudius Regaud - IUCT Oncopole, Toulouse
  - Gustave Roussy, Villejuif